CLINICAL TRIAL: NCT03569176
Title: Superpower Glass Project: A Mobile At-home Intervention for Children With Autism
Brief Title: Examining the Efficacy of a Mobile Therapy for Children With Autism Spectrum Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dennis Paul Wall (Other)
Responsible Party: Sponsor-Investigator, Dennis Paul Wall, Associate Professor, Stanford University
Organization: Stanford University (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-34059
Record Dates: First submitted 2018-06-14; First posted 2018-06-26 (Actual); Results first posted 2024-09-23 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-11

CONDITIONS: Autism Spectrum Disorder
Keywords: mobile health, autism, ASD, mobile therapy, digital, wearable computing, technology
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Autism Glass Intervention (Experimental): Participants in the experimental group will receive the autism glass for 6 weeks once they are assigned to the experimental condition. Participants will be asked to use the glasses at least 3 times a week for 20 minutes sessions in addition to continuing Applied Behavior Analysis (ABA) therapy.
  Interventions: Device: Autism Glass
- Crossover Control for Autism Glass (Other): Participants randomized to the control arm, will continue treatment as usual (receiving ABA twice a week) while the intervention participants will receive the Autism Glass intervention (while continuing to receive ABA therapy). After 6 weeks, control participants will receive the Autism Glass intervention after which, they will be asked to come in for a second round of follow-up testing following 6 weeks of use (at week 18).
  Interventions: Device: Autism Glass

INTERVENTIONS:
Device: Autism Glass — The intervention uses the outward-facing camera on the google glasses to read facial expressions and provides social cues within the child's natural environment during usual social interaction and during games accessed via the smartphone application. Participants who receive the Google Glass intervention will be asked to use it for around 20 minutes 3 times a week with their parents or during ABA therapy.

SUMMARY:
The purpose of this research is to study the effects of a novel artificial intelligence (AI) tool for automatic facial expression recognition that runs on Google Glass through an Android app to deliver social emotion cues to children with autism during social interactions. This novel device will use a camera, microphone, head motion tracker to analyze the behavior of the subject during interactions with other people. The system is designed to give participants non-interruptive social cues in real-time and will record social responses that can later be used to help aid behavioral therapy. It is hypothesized that the system's ability to provide continuous behavioral therapy during social interactions will enable faster gains in social skills.

ELIGIBILITY:
Inclusion Criteria:

1. the child has been diagnosed professionally with ASD
2. the child is currently receiving ABA therapy at least twice per week at home.
3. The child's family is willing to drive to Stanford University for up to 4 study appointments.

Exclusion Criteria:

1. The child scores less than 15 on the Social Communication Questionnaire
2. The child's family does not speak English

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 74 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2018-04-11 (Actual); Study Completion 2018-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis P Wall, PhD, Principal Investigator — Associate Professor

REFERENCES:
- [Derived] Voss C, Schwartz J, Daniels J, Kline A, Haber N, Washington P, Tariq Q, Robinson TN, Desai M, Phillips JM, Feinstein C, Winograd T, Wall DP. Effect of Wearable Digital Intervention for Improving Socialization in Children With Autism Spectrum Disorder: A Randomized Clinical Trial. JAMA Pediatr. 2019 May 1;173(5):446-454. doi: 10.1001/jamapediatrics.2019.0285. PMID 30907929

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: N=3 participants were excluded due to a randomization error.
Period: Baseline (week0) to Post-Test 1 (week6)
Arm/Group | Autism Glass Intervention | Crossover Control for Autism Glass
Started | 40 | 31
Completed | 27 | 25
Not Completed | 13 | 6
Period: Post-Test1(week6) to Post-Test2(week12)
Arm/Group | Autism Glass Intervention | Crossover Control for Autism Glass
Started | 27 | 25
Completed | 24 (Treatment participants completed procedures at Post-test 2 (did not receive Post-Test 3).) | 12
Not Completed | 3 | 13
Period: Post-Test1(week12) to Post-Test2(week18)
Arm/Group | Autism Glass Intervention | Crossover Control for Autism Glass
Started | 0 | 12
Completed | 0 | 12 (Completed at Post-Test 3.)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Autism Glass Intervention | Crossover Control for Autism Glass | Total
Number analyzed (Participants) | 40 | 31 | 71
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.64 (2.52) | 7.94 (1.69) | 8.38 (2.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 37 | 26 | 63
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race and Ethnicity: Caucasian or Euro-American | 12 | 10 | 22
  Race and Ethnicity: African American | 1 | 0 | 1
  Race and Ethnicity: East Asian or Asian American | 9 | 4 | 13
  Race and Ethnicity: South Asian or Indian American | 1 | 4 | 5
  Race and Ethnicity: Middle Eastern or Arab American | 0 | 0 | 0
  Race and Ethnicity: Native American or Alaskan Native | 0 | 0 | 0
  Race and Ethnicity: Hispanic/Latino/Spanish Origin | 7 | 5 | 12
  Race and Ethnicity: More than one race selected | 2 | 6 | 8
  Race and Ethnicity: Unknown/Not Listed | 8 | 2 | 10
Stanford-Binet Intelligence Scales, Abbreviated Battery, Fifth Edition (ABIQ) [Mean (Standard Deviation); unit: points] — The ABIQ assessment measures a child's IQ based on an abbreviated (10 minute) task that measures Nonverbal Fluid Reasoning and Verbal Knowledge to create a standard score for IQ. It will be completed for each child during Intake. The Area Scores and Test Composite on the Stanford-Binet test have an average score of 100 and a standard deviation of 16. The converted score of the individual being assessed indicates where he/she is relative to the norm. A score exceeding 145 is classified as "Genius or near genius," and scores below 70 are classified as "Borderline deficiency."
  points | 75.7 (20.71) | 80.42 (22.61) | 77.76 (21.53)
Mobilized Machine Learning Autism Risk Assessment (MARA) score of autism severity [Mean (Standard Deviation); unit: units on a scale] — The MARA screens for, quantifies, and tracks the severity of core autism symptoms. Parents respond to the survey and it takes less than 5 minutes to complete. The core behavioral domains the MARA focuses on are communication, social reciprocity, and restricted, repetitive, and stereotyped behaviors. Each response to a question is run through a machine learning model that uses an alternating decision tree algorithm to generate a total score ranging from most severe, -10 to least severe, 7.
  units on a scale | -5.57 (4.08) | -4.33 (4.37) | -5.02 (4.22)
Social Communication Questionnaire (SCQ) score [Mean (Standard Deviation); unit: points] — The Social Communication Questionnaire (SCQ) screens for autism in children over 4:0 years in age. Parents are asked 40 Yes/No questions and the resulting score is out of 39 (the first question is not associated with a numerical value). Each item is scored either 1 = presence of abnormal behavior, or 0 = absence of abnormal behavior. Possible scores for verbal children range from 0-39. A score of 15 or above is indicative of autism and is required to be eligible in the research study.
  points | 23.43 (5.13) | 25.06 (4.81) | 24.14 (5.03)

OUTCOME MEASURES:

1. Primary Outcome: Change in Socialization Subscale Scores of the Vineland Adaptive Behavior Scales, 2nd Edition (VABS-II) From Baseline to Week 6.
Description: Vineland Adaptive Behavior Scales, 2nd edition (VABS-II) Socialization subscale will be conducted at the university by a trained research team member. Scores from the socialization domain of the VABS-II reflects one's functioning in social situations. The socialization subscale is 32 items, where raw scores are converted to IQ-type standard scores (mean: 100 sd: 15) for each domain and for the composite adaptive behavior score.The socialization subscale is 32 items, where raw scores are converted to IQ-type standard scores--v-scale scores (M=15, SD=3) where scores range from 1 to 24, and factor in age equivalents, growth scale values, and higher scores indicate better adaptive functioning.
Time Frame: Baseline (week 0), Week 6
Population: Averages at baseline are averages from the original N=40 intervention cohort and N=31 crossover control cohort.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Autism Glass Intervention | Crossover Control for Autism Glass
Number analyzed (Participants) | 40 | 31
score on a scale
  Baseline (week 0) | 68.75 (16.63) | 70.40 (13.26)
  Post-Test 1 (week 6): number analyzed (Participants) | 27 | 25
  Post-Test 1 (week 6) | 71.72 (15.24) | 68.6 (10.80)

2. Primary Outcome: Change in Parent Rated Social Responsiveness Scale 2 (SRS-2) From Baseline to Week 6
Description: The SRS-2 is a 65-item measure where parents rate their child selecting responses on a Likert Scale. This measure will be used to measure and identify social impairment associated with Autism Spectrum Disorder (ASD) and to quantify its severity. Social Responsiveness Scale (SRS) raw scores measure social abilities with lower scores indicating better social skills. (Raw Score Range: 0 - 195 and T-Score Range: 37- above 90).
Time Frame: Baseline (week 0), Week 6
Population: Averages at baseline are averages from the original N=40 intervention cohort and N=31 crossover control cohort.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Autism Glass Intervention | Crossover Control for Autism Glass
Number analyzed (Participants) | 40 | 31
score on a scale
  Baseline (week 0) | 80.68 (8.41) | 80.76 (10.98)
  Post-Test 1 (week 6): number analyzed (Participants) | 27 | 25
  Post-Test 1 (week 6) | 78.4 (8.65) | 81.79 (8.38)

3. Primary Outcome: Change in Emotion Guessing Game (EGG) Scores From Baseline to Week 6
Description: The Emotion Guessing Game is a novel test created for purposes of this study to evaluate the child's ability to correctly label emotions expressed by an examiner in real time. EGG is a pre-set list of 8 emotions, listed 5 times each (Happy, Sad, Angry, Afraid, Surprised, Calm, Disgust, and "Meh"/contempt). During the quick 40-question evaluation, the research coordinator first lists the various emotion choices to the child before beginning the evaluation. Then, the examiner acts out each emotion listed, in order, and waits for a guess from the child, who labels the emotion. The EGG is scored by summing the number of correct responses from the child, higher scores indicated better emotion recognition, where scores can range from 0 to 40.
Time Frame: Baseline (week 0), Week 6
Population: Averages at baseline are averages from the original N=40 intervention cohort and N=31 crossover control cohort.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Autism Glass Intervention | Crossover Control for Autism Glass
Number analyzed (Participants) | 40 | 31
score on a scale
  Baseline (week 0) | 22.80 (11.52) | 24.74 (11.66)
  Post-Test 1 (week 6) | 30.03 (9.44) | 26.88 (11.44)

4. Secondary Outcome: Change in ASD Symptoms as Measured by Brief Observation of Social Communication Change (BOSCC) From Baseline to Week 6
Description: The Brief Observation of Social Communication Change (BOSCC) is designed to measure change in core symptoms of children with autism. It aims to capture change in social communication, interaction, and eye contact. The BOSCC is a play based assessment that consists of two boxes filled with specific toys and takes about 12 minutes to complete.
Time Frame: Baseline (week 0), week 6
Population: While the framework for administration of BOSCC has been published, the scoring algorithm and validation of use in independent replicate samples has not yet been published. Therefore, we were unable to use the BOSCC as initially planned.
Arm/Group | Autism Glass Intervention | Crossover Control for Autism Glass
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change in Adaptive Social and Personal Skills as Measured by Vineland Adaptive Behavior Scales, 2nd Edition (VABS-II) Full Scale From Baseline to Week 6.
Description: The VABS-II is a robust and comprehensive measure of personal and social skills needed in everyday living. The VABS-II covers a child's conceptual, social, and practical skills and can assess children from birth to 90 years. The parent can complete the entire questionnaire in about 20-30 minutes. The raw score in each domain and total raw score are converted to an age-equivalent score. The domain scores are also expressed as standard scores with a mean of 100 and standard deviation of 15. The range for each subscale is from 20 to 140. The subscales are summed to compute a total score, ranging from 80 to 560. The higher the scores are, the better adaptive functioning the children achieve.
Time Frame: Baseline (week 0), week 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Autism Glass Intervention | Crossover Control for Autism Glass
Number analyzed (Participants) | 40 | 31
score on a scale
  Baseline (week 0) | 71.45 (12.66) | 74.63 (10.48)
  Post-Test 1 (week 6) | 72.29 (15.46) | 74.48 (9.79)

6. Secondary Outcome: Change in Child's Emotional, Behavioral, and Social Problems From Baseline (Week 0) to Week 6 as Measured by Child Behavior Checklist (CBCL) Total Score.
Description: The CBCL is a caregiver-directed report that identifies emotional, behavioral, and social problems in children. The patient is rated on 113 items scored on a 3-point Likert-type scale. CBCL total score consists of eight empirically-based syndrome subscales. The total competence score is reported, range: 0-100, where higher scores suggests the more severe symptoms.
Time Frame: Baseline (week 0), Week 6
Population: CBCL Total Score Averages at baseline are averages from the original N=40 intervention cohort and N=31 crossover control cohort.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Autism Glass Intervention | Crossover Control for Autism Glass
Number analyzed (Participants) | 40 | 31
score on a scale
  Baseline (week 0) | 65.95 (7.16) | 69.04 (7.39)
  Post-Test 1 (week 6): number analyzed (Participants) | 27 | 25
  Post-Test 1 (week 6) | 63.77 (6.84) | 65.55 (8.94)

7. Secondary Outcome: Change in NEPSY-II, Affect Recognition Subscale Scores From Baseline to Week 6
Description: The NEPSY-II Affect Recognition subdomain assesses a child's social perception of facial affect recognition. It is designed to assess a child's ability to recognize 6 emotions (happy, sad, angry, fear, disgust, and neutral) from colored photographs of children's faces in four different tasks. Scores range from 1 (well below expected level) to 19 (well above expected level), and have a mean of 10 [standard deviation= 3] that is based on a U.S. normative sample.
Time Frame: Baseline (week 0), Week 6 Baseline (week 0), Week 6 Baseline (week 0), Week 6 Baseline (week 0), week 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Autism Glass Intervention | Crossover Control for Autism Glass
Number analyzed (Participants) | 40 | 31
units on a scale | .099 (.570) | -.068 (.439)

ADVERSE EVENTS:
Time Frame: Participants were assessed over 18-20 weeks.
Arm/Group | Autism Glass Intervention | Crossover Control for Autism Glass
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/31
Other Adverse Events (participants affected / at risk) | 0/40 | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-07): https://cdn.clinicaltrials.gov/large-docs/76/NCT03569176/Prot_SAP_000.pdf